CLINICAL TRIAL: NCT05999760
Title: Retention, Chewing Efficiency and Masticatory Performance of Maxillary Flexible Versus Computer Aided Design/Computer Aided Manufacture(CAD/CAM) Partial Dentures Opposing Fixed Implant Retained Prosthesis.
Brief Title: Retention, Chewing Efficiency and Masticatory Performance of Partial Dentures Opposing Implant Retained Prosthesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Menatallah Mohamed Elhotieby, Principle investigator Researcher fixed and removable prosthodontics, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Elhotieby.M
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Implant Site Reaction; Implant Complication
Keywords: Retention; Chewing efficiency; Removable Prosthodontics

STUDY DESIGN:
Who Masked: Participant
Masking Description: each patient was not informed about material of received prosthesis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (patients received Versacryle removable partial denture) (Active Comparator): patients having Kennedy class I received maxillary Versacryle removable partial denture
  Interventions: Device: evaluation of retention of Versacryle and CAD/CAM partial dentures by force gauge; Device: chewing efficiency by electromyograph(E.M.G); Other: masticatory performance(questionnaire)
- Group II (patients received CAD/CAM fabricated removable partial denture) (Active Comparator): patients having Kennedy class I received maxillary CAD/CAM fabricated removable partial denture
  Interventions: Device: evaluation of retention of Versacryle and CAD/CAM partial dentures by force gauge; Device: chewing efficiency by electromyograph(E.M.G); Other: masticatory performance(questionnaire)

INTERVENTIONS:
Device: evaluation of retention of Versacryle and CAD/CAM partial dentures by force gauge — Evaluation of retention of Versacryle and CAD/CAM partial dentures by force gauge on day one, on first month, and on the second month of prosthesis delivery.
Device: chewing efficiency by electromyograph(E.M.G) — Evaluation of chewing efficiency of Versacryle and CAD/CAM partial dentures by force gauge on day one, on first month, and on the second month of prosthesis delivery.
Other: masticatory performance(questionnaire) — Evaluation of masticatory performance of Versacryle and CAD/CAM partial dentures by questionnaire on day one, on first month, and on the second month of prosthesis delivery.

SUMMARY:
This study aims to evaluate retention ,chewing efficiency and masticatory performance of flexible versus CAD/CAM partial dentures opposing to fixed implant retained restorations.

DETAILED DESCRIPTION:
in this study 22 patients will be selected following inclusion and exclusion criteria. The patients will be divided randomly into two groups.

Group I patients will receive Versacrylic removable partial denture. group II patients will receive CAD/CAM removable partial denture all patients will be given the home care instructions at night and brush cleaning of the dentures.

Measurements of retention using universal testing machine, masticatory performance using T-scan III computerized system and chewing efficiency using chewing function questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker male Patients
* Age ranging from 40-50 years.
* Highly cooperative and motivated patients.
* Patients Systemically free from any immunosuppressive diseases.
* Patients free from Diabetes, Hypertension, Cancer, any mental or physical diseases.
* Patients not receiving any Radiotherapy or chemotherapy treatment.

Exclusion Criteria:

* Female patients
* Smoker patients.
* Age exceeding 50 years
* Uncooperative and unmotivated patients.

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
evaluation of change of retention of versacrylic and CAD/CAM partial denture | on day 1 ,1 month and 2months of prosthesis delivery
  measurement of retention of partial dentures made of Versacryle and CAD/CAM technology
evaluation of change of chewing efficiency of versacrylic and CAD/CAM partial denture | on day 1 ,1 month and 2months of prosthesis delivery
  measurement of chewing efficiency of partial dentures made of Versacryle and CAD/CAM technology
evaluation of change of masticatory performance of versacrylic and CAD/CAM partial denture | on day 1,1 month and 2months of prosthesis delivery
  measurement of masticatory performance of partial dentures made of Versacryle and CAD/CAM technology

CONTACTS AND LOCATIONS:
Overall Officials: Menatallah Elhotieby, Researcher, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Giza, Egypt